CLINICAL TRIAL: NCT00693043
Title: A Pilot Study About Safety and Efficacy of Atomized Intrapleural Lidocaine During Pleuroscopy
Brief Title: Pilot Study About Safety and Efficacy of Atomized Intrapleural Lidocaine During Pleuroscopy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator left the institution requested termination
Sponsor: Lahey Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LCID 2008-007
Record Dates: First submitted 2008-06-02; First posted 2008-06-06 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2014-03

CONDITIONS: Pain
Keywords: Pain control
MeSH Terms: conditions — Pain; Agnosia | interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard anesthesia group (No Intervention): Patients randomized to arm 1 received standard of care anesthesia for pleuroscopy. Duration of the procedure will be recorded. Pain management will be monitored prior to, intraoperatively and at the end of the procedure.
- Lidocaine Group (Experimental): Patients randomized to arm two will receive a reduced topical dose of lidocaine of 2mg/kg and additional lidocaine 3mg/kg infused into the pleura cavity. Duration of procedure will be monitored from the time initial dose of intradermal lidocaine until the start of surgical wound closing, pain scale will be administered prior to the procedure and at the end of the procedure. Lidocaine serum levels will be monitored at 30, 60, and 120 minutes after initial intradermal administration of lidocaine.
  Interventions: Drug: lidocaine hydrochloride

INTERVENTIONS:
Drug: lidocaine hydrochloride — Study group will have up to 2 mg/kg of Lidocaine administered to the skin and additional Lidocaine(3mg/kg)infused through an atomizer using a specialized tip attached to the sterile leur lock syringe into the pleural cavity. The Intrapleural lidocaine dose will be given in a fixed dose of 3 mg/kg. Serum levels will be obtained at 30, 60, and 120 minutes after initial intradermal administration
  Other Names: Drug: lidocaine hydrochloride
  Arms: Lidocaine Group

SUMMARY:
This study will evaluate the potential to decrease the use of IV anesthesia drugs in patients undergoing pleuroscopy administering lidocane standardly applied to the skin in combination with atomized lidocaine applied into the pleural cavity.

DETAILED DESCRIPTION:
Most patient discomfort results from direct manipulation or contact with the parietal pleura during chest tube placement, talc instillation or pleural biopsy. This study intends to use combined IV, intradermal and intrapleural anesthesia during pleuroscopy procedures. Intrapleural atomized lidocaine will be applied directly to the parital pleura. This study will evaluate intravenous anesthesia reduction in subjects treated with intrapleural lidocaine, reduction in total procedure timeby minimizing interruptions due to poor pain control, reduce perioperative pain scores and improve patient comfort nad to determine safety of fixed dosage of 3 mg/kg intrapleural lidocaine given during pleuroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with pleural disease
* Patients undergoing pleuroscopy with talc with or w/o biopsy
* Patients aged 18 - 85
* Patients capable of signing informed consent

Exclusion Criteria:

* Severe congestive heart failure
* Hepatic failure, bilirubin > 2mg/dl, ALT,AST 3XULN
* Prior use Lidocaine in 48 hrs
* Hx SA drug reaction to lidocaine or amide local anesthetics
* Second or third degree heart block (w/o pacemaker)
* Sever sinoatrial block (w/o pacemaker)
* Concurrent treatment with quinidine, flecainide, dsopyramide, procainamide (ClassI antirrhythmic agents)
* Prior use or amiodarone hydrochloride
* systolic BP < 90mmHg
* bradycardia
* accelerated idioventricular rhythm

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Improve pain management in patients undergoing pleuroscopy | pre-procedure and post procedure

SECONDARY OUTCOMES:
Reduction of procedure time Measurement of lidocaine serum levels at 30, 60, 120 | time of procedure will be documented;lidocaine levels monitored throught out

CONTACTS AND LOCATIONS:
Overall Officials: David R Riker, MD, Principal Investigator — Lahey Clinic
Locations (1):
- Lahey Clinic, Burlington, Massachusetts, United States